CLINICAL TRIAL: NCT05964920
Title: Does Human Skeletal Muscle Possess an Epigenetic Memory of Testosterone?
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Adam Sharples, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TESTO-MEM
Record Dates: First submitted 2023-06-16; First posted 2023-07-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy Aging; Age-Related Sarcopenia; Testosterone Deficiency
Keywords: Healthy aging; Preventing Age-related Sarcopenia; Overcoming Anabolic Resistance; Anti-Doping
MeSH Terms: interventions — Sodium Chloride; testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): The placebo group will complete 10-week treatment period where they continue with their regular habitual daily physical activity and receive two placebo (saline) injections (at baseline and week 3). They will then undergo a 12-week period with no treatment and no training, where they just do their regular habitual daily physical activity. Before they undertake a period of structured, progressive resistance training for 10-weeks.
  Questionnaires, physiological and psychological measures, skeletal muscle biopsies and blood samples will be taken at time points of:
  1. Baseline (week 0)
  2. Treatment period (week 10)
  3. Detraining and placebo abstinence (week 22)
  4. Retraining (week 32)
  Interventions: Drug: Saline
- Testosterone Undecanoate (Experimental): The testosterone group will complete 10-week treatment period where they continue with their regular habitual daily physical activity and receive two testosterone undecanoate (Nebido) injections (1000 mg/4 ml at baseline and 500 mg/2 ml week 3). They will then undergo a 12-week period with no treatment and no training, where they just do their regular habitual daily physical activity. Before they undertake a period of structured, progressive resistance training for 10-weeks.
  Questionnaires, physiological and psychological measures, skeletal muscle biopsies and blood samples will be taken at time points of:
  1. Baseline (week 0)
  2. Treatment period (week 10)
  3. Detraining and testosterone abstinence (week 22)
  4. Retraining (week 32)
  Interventions: Drug: Testosterone Undecanoate
- Resistance exercise training + Placebo (Placebo Comparator): The resistance exercise training + placebo group will complete 10-week treatment period where they undergo a period of structured, progressive resistance training and receive two placebo (saline) injections (at baseline and week 3). They will then undergo a 12-week period with no treatment and no training, where they return to their regular habitual daily physical activity. Before they undertake a second period of structured, progressive resistance training for 10-weeks.
  Questionnaires, physiological and psychological measures, skeletal muscle biopsies and blood samples will be taken at time points of:
  1. Baseline (week 0)
  2. Treatment period (week 10)
  3. Detraining and placebo abstinence (week 22)
  4. Retraining (week 32)
  Interventions: Drug: Saline + Resistance exercise training
- Resistance exercise training + Testosterone Undecanoate (Experimental): The resistance exercise training + testosterone group will complete 10-week treatment period where they undergo a period of structured, progressive resistance training and receive two testosterone undecanoate (Nebido) injections (1000 mg/4 ml at baseline and 500 mg/2 ml week 3). They will then undergo a 12-week period with no treatment and no training, where they return to their regular habitual daily physical activity. Before they undertake a second period of structured, progressive resistance training for 10-weeks.
  Questionnaires, physiological and psychological measures, skeletal muscle biopsies and blood samples will be taken at time points of:
  1. Baseline (week 0)
  2. Treatment period (week 10)
  3. Detraining and testosterone abstinence (week 22)
  4. Retraining (week 32)
  Interventions: Drug: Testosterone Undecanoate + Resistance exercise training

INTERVENTIONS:
Drug: Saline — Two placebo injections one at baseline and one week 3.
  Other Names: Placebo
  Arms: Placebo
Drug: Testosterone Undecanoate — Two testosterone undecanoate injections, 1000 mg/4 ml at baseline, 500 mg/2 ml at week 3.
  Other Names: Nebido, Grünenthal (Grünenthal Norway AS)
  Arms: Testosterone Undecanoate
Drug: Saline + Resistance exercise training — Two placebo injections one at baseline and one week 3 and10 weeks of supervised, structured, progressive resistance training.
  Other Names: Placebo + Resistance exercise training
  Arms: Resistance exercise training + Placebo
Drug: Testosterone Undecanoate + Resistance exercise training — Two testosterone undecanoate injections, 1000 mg/4 ml at baseline, 500 mg/2 ml at week 3 and 10 weeks of supervised, structured, progressive resistance training.
  Other Names: Nebido, Grünenthal (Grünenthal Norway AS) + Resistance exercise training
  Arms: Resistance exercise training + Testosterone Undecanoate

SUMMARY:
This project's primary aim of this double-blinded, randomised, placebo-controlled trial is to investigate whether short-term testosterone administration +/- resistance exercise training induces a muscle memory response that can lead to longer-lasting benefits in aged human skeletal muscle.

The investigators will provide older men with the anabolic hormone, testosterone or placebo, with or without resistance training, followed by a period of testosterone abstinence and detraining, followed by a subsequent repeated period of resistance training (retraining). This will help determine if earlier encounters with short-term testosterone administration can be "remembered" and if adaptation to later retraining can be enhanced as a consequence of encountering testosterone earlier.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary males
* 55-70 years old
* Serum testosterone levels >8 nmol/L measured in the morning
* Without any known illness, disease or other conditions
* Undergone screening through medical questionnaire, physical examination, routine blood tests and urine sample
* Written informed consent received

Exclusion Criteria:

* Current or previous participation in a formal exercise regime
* A BMI < 18 or > 30 kg·m2
* Hypersensitivity to the study drug or to any of its constituents
* Active cardiovascular disease: uncontrolled hypertension (BP > 160/100 mmHg), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event
* Family history of early (<55y) death from cardiovascular disease
* Haematocrit >50%
* Malignancy
* Prostate-specific antigen (PSA) >4 ng/mL
* Lower urinary tract symptoms
* Taking beta-adrenergic blocking agents, statins, non-steroidal anti-inflammatory drugs
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial), epilepsy
* Respiratory diseases including: pulmonary hypertension, chronic obstructive pulmanary disease (COPD), asthma, sleep apnoea
* Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, type 1 or 2 diabetes
* Active inflammatory bowel or renal disease
* Current or previous steroid treatment or hormone replacement therapy
* Clotting dysfunction
* Musculoskeletal or neurological disorders
* Alcohol or drug abuse
* Receiving oral anticoagulants
* Serum testosterone levels above the reference range for 50 year olds (>32 nmol/L) (Bjerner et al., 2009) measured in the morning 1

Ages: 55 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Fat-free mass | Baseline and weeks 10, 22, 32
  Change and differences in fat-free mass (g) measured by dual x-ray absorptiometry (DEXA).
Skeletal muscle size and cross-sectional area (CSA) | Baseline and week 5,10, 16, 22, 27, 32
  Change and differences in skeletal muscle size and CSA measured by ultrasound
Skeletal muscle fibre CSA | Baseline and weeks 10, 22, 32
  Change and differences in skeletal muscle fibre CSA measure determined by immunohistochemistry

SECONDARY OUTCOMES:
DNA methylation in skeletal muscle and blood | Baseline and weeks 10, 22, 32
  Methylation measured in difference/fold change values relative to appropriate controls.
Gene expression in skeletal muscle and blood | Baseline and weeks 10, 22, 32
  Gene expression measured in difference/fold change values relative to appropriate controls.
Myonuclei | Baseline and weeks 10, 22, 32
  Change and differences in number of myonuclei determined by immunohistochemistry
Satellite cells | Baseline and weeks 10, 22, 32
  Change and differences in number of satellite cells determined by immunohistochemistry
Isometric muscle strength | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in peak muscle strength (N) using isokinetic dynamometry
Dynamic muscle strength | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in 1-repetition maximum
Muscle force-velocity profiling | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in force (N) and velocity (m/s) derived from a 10-repetition FV-test

OTHER OUTCOMES:
Skeletal muscle stiffness | Baseline and weeks 10, 22, 32
  Change and differences in skeletal muscle stiffness measured by shear wave ultrasonography
Skeletal muscle tissue characteristics | Baseline and weeks 10, 22, 32
  Change and differences in skeletal muscle tissue characteristics determined by immunohistochemistry of muscle biopsies
Bone mineral density | Baseline and weeks 10, 22, 32
  Change and differences in bone mineral density (g/cm2) measured by DEXA
Bone health | Baseline and weeks 10, 22, 32
  Change and differences in bone health determined by bone health biomarkers in blood
Blood volume, haemoglobin and lean body mass | Baseline and weeks 10, 22, 32
  To investigate the association between blood volume, haemoglobin mass and lean body mass measured by carbon monoxide (CO) rebreathing and DEXA.
Blood parameters | Baseline and weeks 10, 22, 32
  Change and differences in steroid hormones in blood (testosterone, androstenediol, estradiol, and other relevant steroid markers, reproductive hormones (LH, FSH), binding protein (SHBG), cholesterol (total cholesterol, LDL, HDL), and PSA level, and endocrine biomarkers (IGF-1 and P-III-NP).
Aging males symptoms | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in Aging male symptoms score (1="none", 5="extremely severe")
Well-being | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in WHO5 well-being index score (0="at not time", 5="all of the time")
Psychological distress | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in SCL-10 symptoms score (1="not at all", 4="extremely")
Fatigue | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in shortened fatigue questionnaire score (1="yes, that is true", 7="no, that is not true")
Sleep | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in Jenkins sleep scale score (0="not at all", 5="22-31days")
Sexual function | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in sexual function score (items from Health-related quality of life (HRQOL) questionnaire), (
Body perception | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in Body Perception Questionnaire very short form score (1=never, 5=always)
Anger | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in The State Anger subscale of STAXI-2score (0="not at all", 3="very much")
Mania | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in Altman Self-Rating Mania Scale (ASRM) score
Suicide thoughts | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in Suicide thoughts from Montgomery and Åsberg Depression Rating Scale
Cognitive function | Baseline and weeks 5, 10, 16, 22, 27, 32
  Change and differences in cognitive function measured by emotion recognition tasks and cognitive reflection tasks
Exercise motivation | Baseline and weekly up to week 10, and weekly from week 22 up to week 32
  Change and differences in perceived motivation score and motivation type
Exercise effort | Baseline and weekly up to week 10, and weekly from week 22 up to week 32
  Change and differences in rating of perceived exertion for effort (Borg CR-10 RPE)
Exercise discomfort | Baseline and weekly up to week 10, and weekly from week 22 up to week 32
  Change and differences in rating of perceived exertion for discomfort (sRPD) score
Session pleasure and displeasure | Baseline and weekly up to week 10, and weekly from week 22 up to week 32
  Change and differences in perceived pleasure/displeasure with the training session using the pleasure/displeasure feeling scale (sPDF), (-5=very bad", 5="very good")
Exercise enjoyment | Baseline and weekly up to week 10, and weekly from week 22 up to week 32
  Change and differences in exercise enjoyment scale score (1="not at all", 7=extraordinary")
Reps in reserve | Baseline and weekly up to week 10, and weekly from week 22 up to week 32
  Change and differences in the ability to predict reps in reserve

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No identifiable information will be included in any publication. Genome-Wide DNA Methylation and Gene Expression will be deposited with full open access on Gene Expression Omnibus (GEO) (https://www.ncbi.nlm.nih.gov/geo/) an internationally recognised database. GEO data derived from human samples will be anonymous, with no identifiable information. GEO data will be deposited at the same time as a publication. All non-identifiable results from the project will be ultimately published in peer-reviewed journals. In addition, all image files, raw excel/ .csv / txt /word files for any of the other analyses described above in the methods will be available as either supplementary files on the publisher's website or fully accessible on request to the corresponding author/authors.

REFERENCES:
- [Background] Egner IM, Bruusgaard JC, Eftestol E, Gundersen K. A cellular memory mechanism aids overload hypertrophy in muscle long after an episodic exposure to anabolic steroids. J Physiol. 2013 Dec 15;591(24):6221-30. doi: 10.1113/jphysiol.2013.264457. Epub 2013 Oct 28. PMID 24167222
- [Background] Seaborne RA, Strauss J, Cocks M, Shepherd S, O'Brien TD, van Someren KA, Bell PG, Murgatroyd C, Morton JP, Stewart CE, Sharples AP. Human Skeletal Muscle Possesses an Epigenetic Memory of Hypertrophy. Sci Rep. 2018 Jan 30;8(1):1898. doi: 10.1038/s41598-018-20287-3. PMID 29382913
- [Background] Turner DC, Seaborne RA, Sharples AP. Comparative Transcriptome and Methylome Analysis in Human Skeletal Muscle Anabolism, Hypertrophy and Epigenetic Memory. Sci Rep. 2019 Mar 12;9(1):4251. doi: 10.1038/s41598-019-40787-0. PMID 30862794
- [Background] Sharples AP, Turner DC. Skeletal muscle memory. Am J Physiol Cell Physiol. 2023 Jun 1;324(6):C1274-C1294. doi: 10.1152/ajpcell.00099.2023. Epub 2023 May 8. PMID 37154489
- [Background] Gharahdaghi N, Rudrappa S, Brook MS, Idris I, Crossland H, Hamrock C, Abdul Aziz MH, Kadi F, Tarum J, Greenhaff PL, Constantin-Teodosiu D, Cegielski J, Phillips BE, Wilkinson DJ, Szewczyk NJ, Smith K, Atherton PJ. Testosterone therapy induces molecular programming augmenting physiological adaptations to resistance exercise in older men. J Cachexia Sarcopenia Muscle. 2019 Dec;10(6):1276-1294. doi: 10.1002/jcsm.12472. Epub 2019 Sep 30. PMID 31568675
- [Background] Sharples AP, Polydorou I, Hughes DC, Owens DJ, Hughes TM, Stewart CE. Skeletal muscle cells possess a 'memory' of acute early life TNF-alpha exposure: role of epigenetic adaptation. Biogerontology. 2016 Jun;17(3):603-17. doi: 10.1007/s10522-015-9604-x. Epub 2015 Sep 8. PMID 26349924
- [Background] Wen Y, Dungan CM, Mobley CB, Valentino T, von Walden F, Murach KA. Nucleus Type-Specific DNA Methylomics Reveals Epigenetic "Memory" of Prior Adaptation in Skeletal Muscle. Function (Oxf). 2021 Aug 5;2(5):zqab038. doi: 10.1093/function/zqab038. eCollection 2021. PMID 34870208